CLINICAL TRIAL: NCT03928119
Title: Construction of Modern reGional Network for Acute Myocardial Infarction
Brief Title: reGional Network for Acute Myocardial Infarction
Acronym: GAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Maoming People's Hospital (Other); Dongguan People's Hospital (Other Government); Southern Medical University, China (Other); Guangzhou Panyu Central Hospital (Other); Yangjiang People's Hospital (Other); Shenzhen People's Hospital (Other); Longyan First Hospital, Affiliated to Fujian Medical University (Unknown)
Responsible Party: Principal Investigator, Jiyan Chen, Professor, Guangdong Provincial People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014B070706010
Record Dates: First submitted 2019-04-21; First posted 2019-04-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Coronary Heart Disease; Acute Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction
Keywords: Acute myocardial infarction; STEMI; regional network
MeSH Terms: conditions — Coronary Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): community public education, non-PCI center and emergency transfer system improvement, and inhospital green-channal optimization for PCI center.
  Interventions: Behavioral: public education and network construction
- Control group (No Intervention): Usual care of AMI public and medical health service

INTERVENTIONS:
Behavioral: public education and network construction — Publication education includes multiple methods of acute myocardial infarction knowledge education. Network construction includes regional connection of ST-Segment Elevation Myocardial Infarction patients transfer for percutaneous coronary intervention treatment, as well as physicians skill improvement in primary hospital.
  Arms: Intervention group

SUMMARY:
Incidence of ST-segment Elevation Myocardial Infarction (STEMI) is rising and the existing emergency medical aid system for STEMI was not enough for timely perfusion treatment. No existing research with high-quality data focuses on the characteristic of STEMI incidence and regional network construction. Aiming of Guangdong GAMI(reGional network for Acute Myocardial Infarction) project is to establish effective collaborative regional network system for STEMI patients treatment.

DETAILED DESCRIPTION:
The project of Guangdong GAMI(reGional network for Acute Myocardial Infarction) is being conducted during 2015-2019 in eight districts with diverse economic development across southern China (Integrated care model was conducted in four regions, which mainly included community public education, non primary-PCI capable centre and referral system improvement, and inhospital green-channal optimization for primary-PCI capable centre. Other four centers were underwent usual care of acute myocardial infacrtion public and medical health service). All the ST-segment elevation myocardial infarction (STEMI) patients admitted in the hospital within 30 days from the symptom onset were enrolled. The key data of the timeline of STEMI onset and treatment were precisely recorded. Other details of STEMI treatment in hospitals such as laboratory data and medication were also collected. During the research period, actions of both optimizing the regional STEMI patients transfer and treatment to shorten the medical delay, as well as educating the public to improve their awareness of early treatment of STEMI were taken meanwhile. In addition, laboratory data, medication, and follow-up information were recorded in a database for further analysis regarding the STEMI patient treatment.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who suspected diagnosis with STEMI.

Exclusion Criteria:

1. patients refused to undergo coronary angiography;
2. patients were confirmed as non-STEMI by coronary angiography or the course of STEMI over 1 month;
3. patients occurred onset STEMI during hospitalization in hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7102 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Receipt of reperfusion therapy within 12 hoursInfarction patients | From 1 month before hospitalization to 24 hours after hospitalization
  The primary outcome was the proportion of patients who received symptom-to-reperfusion treatment within 12 hours.

SECONDARY OUTCOMES:
Onset-to-admission time within 12 hours | From 1 month before hospitalization to 24 hours after hospitalization
  The proportion of patients who take a symptom-to-admission period within 12 hours.
Door-to-balloon time within 90 minutes | 24 hours
  The proportion of patients who take a door-to-balloon period within 90 minutes.
In-hospital clinical outcomes | 30 days
  The incidence of several in-hospital outcomes (in-hospital death; and major adverse cardiac events [MACEs], which mainly included in-hospital death, recurrence of myocardial infarction, and stroke); the length of stay.
1-year all-cause mortality | 1 year
  Total mortality between 30 days and 1 year after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liang, MD, Principal Investigator — Maoming People's Hospital; Jianfeng Ye, MD, Principal Investigator — Dongguan People's Hospital; Yunzhao Hu, MD, Principal Investigator — The first People's Hospital of Shunde, Foshan; Wenzhu Zhang, MD, Principal Investigator — Guangzhou Panyu Central Hospital
Locations (8):
- China (8):
  - Longyan First Hospital Affiliated to Fujian Medical University, Longyan, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - People's Hospital of Yangjiang, Yangjiang, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu J, Xuan S, Downing NS, Wu C, Li L, Krumholz HM, Jiang L. Protocol for the China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Million Persons Project pilot. BMJ Open. 2016 Jan 4;6(1):e010200. doi: 10.1136/bmjopen-2015-010200. PMID 26729395
- [Background] Yin X, He Y, Zhang J, Song F, Liu J, Sun G, Liang Y, Ye J, Hu Y, Song M, Chen C, Xu Q, Tan N, Chen J, Liu Y, Liu H, Tian M. Patient-level and system-level barriers associated with treatment delays for ST elevation myocardial infarction in China. Heart. 2020 Oct;106(19):1477-1482. doi: 10.1136/heartjnl-2020-316621. Epub 2020 Jun 24. PMID 32580976
- [Derived] Liu Y, Liu J, Liang Y, Ye J, Hu Y, Chen L, Dong S, Huang X, Song M, Meng R, Zheng X, He Y, Zhang J, Yin X, Chen S, Tan N, Tian M, Chen J. Effect of an integrated care model on ST-segment elevation myocardial infarction management in China: a prospective, multicentre, non-randomised controlled study. Heart. 2025 Sep 9:heartjnl-2024-324155. doi: 10.1136/heartjnl-2024-324155. Online ahead of print. PMID 40930595